CLINICAL TRIAL: NCT03053778
Title: Individualised Follow-up After Valve Surgery
Acronym: INVOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Britt Borregaard, Principal Investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 222
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Heart Valve Diseases; Surgery; Readmission
Keywords: Readmission; Early follow-up; Heart valves; Heart valve surgery
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Early follow-up after discharge
  Interventions: Other: Early follow-up

INTERVENTIONS:
Other: Early follow-up — Early follow-up until 4 weeks after discharge

SUMMARY:
This study aims to investigate the effect of an intervention consisting of early, individualised outpatient follow-up after heart valve surgery on unplanned readmissions and death within 180-days after discharge.

Furthermore, Health economics and health-related quality of life will be investigated.

DETAILED DESCRIPTION:
The incidence of valvular heart disease is estimated to exceed 42 million people worldwide. In Denmark 1700 patients undergo heart valve surgery every year and the number is increasing due to an ageing population. The most common heart valve diseases is aortic stenosis, followed by mitral regurgitation and aortic regurgitation, whereas only few patients are treated in Denmark for mitral stenosis and primary tricuspid valve and pulmonic valve diseases.

Heart valve surgery can be a lifesaving procedure for patients with severe symptomatic heart valve disease, but complications after heart valve surgery are common and readmissions frequent with rates exceeding 40% in Denmark. Most frequent causes for readmission, includes new onset atrial fibrillation, pleural and pericardial effusions, infections and acute heart failure. These causes can potentially be detected by careful outpatient follow-up in order to avoid unplanned readmission, and improve mental, physical and social health outcomes. A recent Danish study demonstrated that 56% of surgical heart valve patients were readmitted within a year and readmission was associated with low psychical and mental PROs. PROs' include validated patient health status surveys that allow quantification of critical patient-centered outcomes. Further previous studies have suggested an association between PROs and prolonged hospital stay, morbidity and mortality in cardiac patients. Knowledge about PROs can potentially be used to identify patients that especially may benefit from intensified follow-up after heart valve surgery.

Existing guidelines recommend that patients following valve surgery are reviewed on a regular basis by a cardiologist with special knowledge about heart valve diseases. A recent European study demonstrate though, a gap between the existing guidelines and clinical practice. A plausible way to improving the postoperative care could be to introduce a multidisciplinary heart valve clinic (HVC), where specialized nurses educates the patients while intervening and supporting the patients after surgery in collaboration with cardiologist and surgeons. This has proven efficient in improving outcomes such as, mortality, readmission and quality of life in patients with heart failure.3 A multidisciplinary teamwork can provide a timely access to a clinical review of the patient and simultaneously look for signs and symptoms of valve dysfunction.18 Although, previous studies have described the HVCs. Although, previous studies have described the HVCs, the effect gained from HVC compared to usual care on readmission, mortality, cost-utility and patient-reported outcomes have not yet systematically been investigated.

The aim for this study is firstly to describe PROs after heart valve surgery, incorporate the knowledge into a structured intervention, and secondly to evaluate a HVC and its association to PRO's, readmission, mortality and cost-utility.

The study consist of two parts,

* Matched cohort study comparing HVC to a historical control group to evaluate the effect of the HVC on readmission, mortality and HRQoL.
* A health economic analysis of effect of the HVC compared to a historical control Group.

The intervention and collection of clinical data: Introducing a HVC to gain knowledge of its effect on readmission, mortality and health economics.

Preoperative: Clinical data regarding the patient will be gathered at admission including calculated Euroscore II, pulmonary function measured with spirometry, status on nutrition, smoking and alcohol consumption, BMI, electrocardiography (ECG), and most recent echocardiography. Furthermore, the patients' frailty status will be assessed with a gait speed test the day before surgery and will be used in the risk model.

Postoperative: Before discharge a trained cardiac nurse will perform a screening for pleural and pericardial effusion, volume overload, risk for atrial fibrillation and repeat frailty assessment. Before discharge the patients' medication will be evaluated and adapted according to their clinical status, and the patients will be educated in warning signs after surgery. The surgical status will be evaluated before discharge. Based on these data and the PROs the patients' follow-up will be individualized.

Follow-up: The specific follow-up will be planed according to the patients' status where patients considered at high risk of being readmitted based on the clinical evaluation at discharge (e.g. atrial fibrillation) will have a more intensive follow-up. The focus of the follow-up will be a status on the patients' physical condition regarding; weight, pain and shortness of breath in combination with the areas of the PROs from study I. Consideration on further follow-up will be made depending on the condition of the patient.

After 1 month all patients will be seen in the HVC where ECG and echocardiography will be performed. At each visit the patient will be educated and informed regarding the disease and illnesses, which should lead to a better understanding and self-management of care in the post-operative period. The aim of the education is to give the patient the insight to promptly identify and report the symptoms and signs for progression of their valve disease or dysfunction of their prosthetic or repaired valve. The patient education thereby also aims to improve the patients' wellbeing and psychological condition by an increase of the feeling of security and by preventing poor physical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient having Heart Valve Surgery at Odense University Hospital, Denmark

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Reduction of readmission | Up to two years
  Reduction of readmission. a controlled prospective intervention trial comparing readmission rates and all-cause mortality in patients undergoing individualized follow-up with a historical control Group. A propensity matching will be performed

SECONDARY OUTCOMES:
Differences in costs between the two groups | Up to three years
  Health economics as measured by differences in the two groups. Further more a cost-utility analysis of cost and quality of life. The cost utility analysis is measured with a questionnaire
Quality of Life and associations with readmission | Up to three years
  Symptoms of health related quality of life measured with a questionnaire
The effect of a Heart valve Clinic on patient-reported outcomes | Up to three years
  Symptoms of disease specific quality of life measured with a questionnaire
Frailty status after Heart valve surgery | Up to two years
  Measuring of frailty status at discharge and associations to other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Britt Borregaard, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided